CLINICAL TRIAL: NCT02886065
Title: A Phase 1b Study of PVX-410, a Multi-Peptide Cancer Vaccine, and Citarinostat (CC-96241), a Histone Deacetylase Inhibitor (HDAC) With and Without Lenalidomide for Patients With Smoldering Multiple Myeloma
Brief Title: A Study of PVX-410, a Cancer Vaccine, and Citarinostat +/- Lenalidomide for Smoldering MM
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Celgene (Industry); OncoPep, Inc. (Industry)
Responsible Party: Principal Investigator, Noopur Raje, MD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-237
Record Dates: First submitted 2016-08-28; First posted 2016-09-01 (Estimated); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Smoldering Multiple Myeloma
Keywords: Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma; Neoplasms, Plasma Cell | interventions — poly ICLC; citarinostat; Lenalidomide; PVX-410 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PVX-410 + Citarinostat (Experimental): Participants will receive:
  * 6 biweekly doses of PVX-410
  * 6 biweekly doses of Hiltonol
  * 3 monthly cycles of Citarinostat
  Interventions: Drug: Hiltonol; Drug: Citarinostat; Biological: PVX-410
- PVX-410 + Citarinostat + Lenalidomide (Experimental): Participants will receive:
  * 6 biweekly doses of PVX-410
  * 6 biweekly doses of Hiltonol
  * 3 monthly cycles of Citarinostat
  * 3 monthly cycles of Lenalidomide
  Interventions: Drug: Hiltonol; Drug: Citarinostat; Drug: Lenalidomide; Biological: PVX-410

INTERVENTIONS:
Drug: Hiltonol — Intramuscular injection of Hiltonol (1 mg) administered Biweekly at the time of PVX-410 administration
  Other Names: Poly ICLC
Drug: Citarinostat — Citarinostat (180 mg) administered orally once daily on days 1-21 every 28 day cycle.
  Other Names: CC-96241
Drug: Lenalidomide — Lenalidomide (25 mg) administered orally once daily on days 1-21 every 28 day cycle.
  Other Names: REVLIMID
  Arms: PVX-410 + Citarinostat + Lenalidomide
Biological: PVX-410 — PVX-410 Biweekly (0.8 mg) via subcutaneous injection

SUMMARY:
This research study is studying a targeted therapy as a possible treatment for Smoldering Multiple Myeloma.

The following intervention will be involved in this study:

* Lenalidomide
* Citarinostat (CC-96241)
* PVX-410

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied.

In this research study, the investigators are studying Smoldering Multiple Myeloma. Smoldering Multiple Myeloma is an early precursor to a rare blood cancer known as Multiple Myeloma, which affects plasma cells. The study will test two different combinations of the study drugs; a combination of the vaccine (PVX-410) along with Citarinostat (CC-96241) and triple combination of the vaccine, Citarinostat, and Lenalidomide.

The vaccine (PVX-410) is a multi-peptide vaccine that contains four synthetic peptides that together are intended to induce a T cell-mediated immune response against the myeloma. The FDA (the U.S. Food and Drug Administration) has not approved PVX-410 as a treatment for any disease.

Citarinostat is an orally active, small-molecule Histone Deacetylase (HDAC) Inhibitor which is being combined here to further augment the immune activity of the vaccine. Citarinostat has not been approved by the FDA as a treatment for any disease.

Lenalidomide is commercially available analogue of thalidomide with immunomodulatory, antiangiogenic, and antineoplastic properties that has demonstrated an increase in immune activity in previous trials. The FDA has approved Lenalidomide as a treatment option for Smoldering Multiple Myeloma. Lenalidomide is being added to the combination of the vaccine and Citarinostat because it is hypothesized that co-administration of lenalidomide along with Citarinostat would further enhance the T cell-mediated immune response induced by PVX-410.

ELIGIBILITY:
Inclusion Criteria:

* Patient has confirmed SMM according to a definition derived from the International Myeloma Working Group (IMWG) definition (International Working Group, 2003): serum M-protein ≥3 g/dL or BMPC >10%, or both, along with normal organ and marrow function (CRAB) within 4 weeks before baseline.

  * C: Absence of hypercalcemia, evidenced by a calcium <10.5 mg/dL.
  * R: Absence of renal failure, evidenced by a creatinine < 1.5 mg/dL (177 µmol/L) or calculated creatinine clearance (using the Modification of Diet in Renal Disease [MDRD] formula) >50 mL/min.
  * A: Absence of anemia, evidenced by a hemoglobin >10 g/dL.
  * B: Absence of lytic bone lesions on standard skeletal survey.
* Patient is at higher than average risk of progression to active MM, defined as having 2 or more of the following features:

  * Serum M-protein ≥3 g/dL.
  * BMPC >10%.
  * Abnormal serum FLC ratio (0.26-1.65).
* Patient is aged 18 years or older.
* Patient has a life expectancy of greater than 6 months.
* Patient is HLA-A2+
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patient has adequate bone marrow function, evidenced by a platelet count ≥75×109/L and an absolute neutrophil count (ANC) ≥1.0×109/L within 2 weeks before baseline.
* Patient has adequate hepatic function, evidenced by a bilirubin ≤2.0 mg/dL and an alanine transaminase (ALT), and aspartate transaminase (AST) ≤2.5×ULN within 2 weeks before baseline.
* If of child-bearing potential, patient agrees to use adequate birth control measures during study participation.
* If a female of child-bearing potential , patient has negative serum pregnancy test results within 2 weeks before baseline and is not lactating.
* If assigned to receive lenalidomide and a female of reproductive potential, must adhere to the scheduled pregnancy testing as required in the Revlimid REMS® program.
* If assigned to receive lenalidomide, patient must be registered into the mandatory Revlimid REMS® program and be willing and able to comply with the requirements of the REMS® program.
* Patient (or his or her legally accepted representative) has provided written informed consent to participate in the study.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Patient has symptomatic MM, as defined by any of the following:

  * Lytic lesions or pathologic fractures.
  * Anemia (hemoglobin <10 g/dL).
  * Hypercalcemia (corrected serum calcium > 11.5 mg/dL).
  * Renal insufficiency (creatinine > 1.5 mg/dL).
  * Other: symptomatic hyperviscosity, amyloidosis.
* Patient has a history of a prior malignancy within the past 3 years (excluding resected basal cell carcinoma of the skin or in situ cervical cancer).
* Patient has abnormal cardiac status, evidenced by any of the following:

  * New York Heart Association (NYHA) stage III or IV congestive heart failure (CHF).
  * Myocardial infarction within the previous 6 months.
  * Symptomatic cardiac arrhythmia requiring treatment or persisting despite treatment.
* Patient is receiving any other investigational agent.
* Patient has a current active infectious disease or positive serology for human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B virus (HBV), or hepatitis A virus (HAV).
* Patient has a history of or current auto-immune disease.
* Patient has been vaccinated with live attenuated vaccines within 4 weeks before study vaccination.
* Any previous treatment with a HDAC inhibitor, including Citarinostat.
* Had involvement in the planning and/or conduct of the study by association with the Sponsor, study drug supplier(s) or study center or was previously enrolled in the present study.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of treatment, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Frediricia's Correction.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, active peptic ulcer disease or gastritis, active bleeding diatheses, or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Safety And Tolerability Of The PVX-410 Tumor Vaccine Regimen | 2 years
  The proportion of participants who experience dose limiting toxicities and other toxicities. The CTCAE version 4 criteria will be used to grade adverse events.

SECONDARY OUTCOMES:
Immune Responses Of Lymphocytes To HLA A2+ | 2 years
Change In Monoclonal (M) Serum Protein | 2 years
Change In Free Light Chain (FLC) | 2 years
Change In Urinary FLC Level | 2 years
Correlation of Immune Response and Clinical Anti-tumor Responses | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Noopur Raje, MD, Principal Investigator — Massachusetts General Hospital
Locations (6):
- United States (6):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospital of Cleveland- Seidman Cancer Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No